CLINICAL TRIAL: NCT03414554
Title: Risk of Hepatocellular Carcinoma in HCV Cirrhotic Patients Treated With Direct Acting Antiviral Drugs.
Brief Title: Risk of HCC in Cirrhotic Patients Post DAAs Ttt
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alshaimaa Mohammed Rafat Ali, Principal investigator at Tropical medicine and Gastroenterology Department, Assiut University
Other Study IDs: HCCDAAs
Record Dates: First submitted 2018-01-23; First posted 2018-01-30 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: HCC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HCV patients receiving DAAs: Patients with HCV-related liver cirrhosis (eligible for treatment) who will recieve DAAs therapy with one year follow up.markers: miR121, miR122, miR124will be assessed in both groups before and after DAAs

SUMMARY:
Direct acting antivirals (DAAs) are a novel and completely oral hepatitis C therapy . DAAs are used in most patients being treated for hepatitis C, including those with decompensated cirrhosis. This type of treatment has now completely replaced interferon-based therapy .Therapy of chronic hepatitis C with direct-acting antivirals (DAAs) is able to induce a sustained virological response (SVR) in over 85% of patients, even if liver cirrhosis is present. Cirrhotic patients should be closely monitored after treatment.HCC is thought to develop over time as the liver is exposed to inflammation and develops fibrosis. Thus, if DAAs can eliminate inflammation mediated by HCV, the risk of HCC should decrease. However, several centers have observed that this actually may not be the case. Tumor genesis occurs through a multistep, multifactorial process. Eliminating HCV-induced inflammation may not be enough to decrease risk of HCC.DAAs have provided an effective, well tolerated treatment for hepatitis C in patents with cirrhosis . However, several studies have shown unexpectedly high rates of recurrence of HCC in the early post DAAs treatment time period.

1. Evalution of occurrence and risk factors for hepatocellular carcinoma (HCC) in patients with HCV-related liver cirrhosis after direct acting antiviral drugs (DAAs) therapy.
2. To asses diagnostic value of novel markers in patients who developed hepatocellular carcinoma (HCC) after (DAAs)

DETAILED DESCRIPTION:
HCV is a worldwide infection, it is estimated that about at about 3.0% (170-200 million people) of the world's population are infected. HCV is associated with an increased disease burden due to liver cirrhosis and considerable mortality . More than 350,000 people dying each year from hepatitis C-related liver disease. Adding to the problem of HCV infection is the presence of occult HCV infection.

Egypt has the highest prevalence worldwide, it is estimated to be 14.7% among a representative sample of Egyptian population, aged 15-59 year . Egypt is among countries responsible for 80.0% of global infections. Further, prevalence is higher among hospitalized patients and special clinical populations.

Hepatitis C virus (HCV) has great genetic variability, with 6 major genotypes (GTs); GT-1 to 6. In Egypt, HCV is almost exclusive GT-4 distribution. HCV has significant differences in their global distribution and prevalence.

Worldwide, Hepatocellular carcinoma (HCC) is the fifth most common cancer in men and the seventh in women. Hepatocellular carcinoma (HCC) is the third leading cause of cancer-related death worldwide and one of the leading causes of death among patients with cirrhosis. In Egypt, HCC is the second most common cancer in men and the sixth most common cancer in women.

Direct acting antivirals (DAAs) are a novel and completely oral hepatitis C therapy . DAAs are used in most patients being treated for hepatitis C, including those with decompensated cirrhosis. This type of treatment has now completely replaced interferon-based therapy .Therapy of chronic hepatitis C with direct-acting antivirals (DAAs) is able to induce a sustained virological response (SVR) in over 85% of patients, even if liver cirrhosis is present. Cirrhotic patients should be closely monitored after treatment.

HCC is thought to develop over time as the liver is exposed to inflammation and develops fibrosis. Thus, if DAAs can eliminate inflammation mediated by HCV, the risk of HCC should decrease. However, several centers have observed that this actually may not be the case. Tumor genesis occurs through a multistep, multifactorial process. Eliminating HCV-induced inflammation may not be enough to decrease risk of HCC.

DAAs have provided an effective, well tolerated treatment for hepatitis C in patents with cirrhosis. However, several studies have shown unexpectedly high rates of recurrence of HCC in the early post DAAs treatment time period.

MicroRNAs (miRNAs) are a set of small, single-stranded, non-coding RNA molecules (21-30 nucleotides) that negatively regulate gene expression at the posttranscriptional level by translational inhibition or degradation of target mRNA, depending on the degree of complementary base pairing. Aberrant expression of miRNA is common in various human malignancies and modulates cancer-associated genomic regions or fragile sites. As for the relationship between miRNA and HCC several studies have demonstrated that the aberrant expression of specific miRNA can be detected in HCC cells and tissues. However, little is known about the mechanisms of miRNA-related cell proliferation and development.ref

Aim of work:

1. Evalution of occurrence and risk factors for hepatocellular carcinoma (HCC) in patients with HCV-related liver cirrhosis after direct acting antiviral drugs (DAAs) therapy.
2. To asses diagnostic value of novel markers in patients who developed hepatocellular carcinoma (HCC) after direct acting antiviral drugs -DAAs -therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HCV-related liver cirrhosis (eligible for treatment) who developed (HCC) after DAAs therapy within one year follow up.
* Age and sex matched group of patients with HCV- related liver cirrhosis who didn't develop HCC after DAAs therapy within one year follow up(as control group)
* Patients with chronic HCV related liver cirrhosis complicated by hepatocellular carcinoma not eligible for treatment.(discovered during enrollment in HCV treatment program)

Exclusion Criteria:

* Patients who refuse to participate in the study.
* Patients with hepatitis B virus, any other causes of cirrhosis.(Alcohol consumpation, Biliary, Cardiac…..etc)
* Patients with cancers other than HCC or metastatic liver cancer.
* Patients who developed HCC on transplanted liver.
* Patients who previously treated for HCC.
* Patients who receive any immunosuppression drugs.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study is a prospective study that will be carried out on patients with HCV-related liver cirrhosis treated with direct acting antiviral drugs at ALRAJHI Liver hospital, Assiut university from February 2018 to December 2019.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-02-01 (Estimated); Primary Completion 2018-12-30 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
Occurrence and risk factors for HCC post DAAs | One year
  Perecentage of occurrence of hepatocellular carcinoma (HCC) in patients with HCV-related liver cirrhosis after direct acting antiviral drugs (DAAs) therapy.

SECONDARY OUTCOMES:
Diagnostic value of miRNA in patients who developed HCC post DAAs | One Year
  Measuring miRNA in patients who developed HCC post DAAs in mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Alshaimaa Rafat, MD, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wartelle-Bladou C, Le Folgoc G, Bourliere M, Lecomte L. Hepatitis C therapy in non-genotype 1 patients: the near future. J Viral Hepat. 2012 Aug;19(8):525-36. doi: 10.1111/j.1365-2893.2012.01634.x. PMID 22762136
- [Background] Xu J, Wu C, Che X, Wang L, Yu D, Zhang T, Huang L, Li H, Tan W, Wang C, Lin D. Circulating microRNAs, miR-21, miR-122, and miR-223, in patients with hepatocellular carcinoma or chronic hepatitis. Mol Carcinog. 2011 Feb;50(2):136-42. doi: 10.1002/mc.20712. Epub 2010 Dec 10. PMID 21229610
- [Background] Pawlotsky JM, Feld JJ, Zeuzem S, Hoofnagle JH. From non-A, non-B hepatitis to hepatitis C virus cure. J Hepatol. 2015 Apr;62(1 Suppl):S87-99. doi: 10.1016/j.jhep.2015.02.006. PMID 25920094
- [Background] Omar A, Abou-Alfa GK, Khairy A, Omar H. Risk factors for developing hepatocellular carcinoma in Egypt. Chin Clin Oncol. 2013 Dec;2(4):43. doi: 10.3978/j.issn.2304-3865.2013.11.07. PMID 25841922
- [Background] Lavanchy D. Evolving epidemiology of hepatitis C virus. Clin Microbiol Infect. 2011 Feb;17(2):107-15. doi: 10.1111/j.1469-0691.2010.03432.x. PMID 21091831